CLINICAL TRIAL: NCT03619980
Title: Retrospective Study to Evaluate Time to Event and Treatment of Prostate Cancer Patients Throughout the Disease States, From m1HSPC and m1CRPC Until Progression or Death.
Brief Title: A Non-Interventional Study to Evaluate Time to Event and Healthcare Resource Utilisation for Prostate Cancer Participants Throughout the Disease Trajectories Until Progression or Death
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 9785-MA-3167; 9785-MA-3631 (Other: Amendment 2 to main study 9785-MA-3167)
Record Dates: First submitted 2018-08-02; First posted 2018-08-08 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Non interventional; Registry
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 11 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with prostate cancer: This is a retrospective registry based study to collect real world data on participants with different disease stages of prostate cancer in Sweden.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Retrospective study to evaluate time to event and healthcare resource utilisation of prostate cancer patients throughout the different disease stages, until progression or death.

SUMMARY:
Primary objective of this study is to describe the time in each prostate cancer stage from non-metastatic Hormone Sensitive Prostate Cancer (m0HSPC), metastatic Hormone Sensitive Prostate Cancer (m1HSPC), non-metastatic Castrate-Resistant Prostate Cancer (m0CRPC), metastatic Castrate-Resistant Prostate Cancer (m1CRPC) to progression or death.

The secondary objectives of this study are to describe co-medication at each disease stage, to describe co-morbidities at each disease stage and to describe the healthcare resource use and costs associated to each disease stage.

This study has been opened and amended (amendment 2; also known as 9785-MA-3631 study) to describe the time in each prostate cancer state from m1HSPC to progression or death. The secondary objective for amendment 2 is to describe co-medication at each disease state, describe co-morbidities at each disease state, and describe PCa treatments in the m1HSPC state. The aim of the second amendment is to provide up to date real world data on the change of the treatment landscape in the m1HSPC population from 1 January 2021 to 30 June 2024.

DETAILED DESCRIPTION:
This is a retrospective analysis of Prostate Cancer patients from m0HSPC, m1HSPC, m0CRPC, m1CRPC followed in the Prostate Cancer Database Sweden (PCBaSe) database. The patient population consists of men recorded in Patient-overview Prostate Cancer (PPC) between 1 January 2014 until death or 31 December 2016. Patient history to 2006 was collected by retrospective charted review.

Data will be extracted from PPC for the different Prostate Cancer (PCa) disease stages, from m0HSPC, m1HSPC, m0CRPC, m1CRPC until progression or death. The prostate cancer disease progression from m0HSPC, m1HSPC, m0CRPC, m1CRPC until progression or death has not been recorded in a systematic way. Given the complexity of this disease, the aim of this study is to have a comprehensive understanding about the disease progression in prostate cancer, from m0HSPC, m1HSPC, m0CRPC, m1CRPC until progression or death.

In addition, the following will be collected: co-morbidities, co-medication, health care resource utilization and costs, as well as other health economic variables such as sick leave and early retirement at the different disease stages.

ELIGIBILITY:
Inclusion Criteria:

* All patients registered in PPC.

Exclusion Criteria:

* None.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with prostate cancer registered in PPC.
Sampling Method: Non-Probability Sample
Enrollment: 6908 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Time from entry to exit either by progression or death from prostate cancer stage m0HSPC | 11 years
  M0HSPC as defined by date for start of ADT (Androgen Deprivation Therapy) (bicalutamide or hormone therapy) and no date for metastatic disease.
Measure: Time from entry to exit either by progression or death from prostate cancer stage m1HSPC | 11 years
  M1HSPC as defined by date for start of ADT (bicalutamide or hormone therapy) and date for metastatic disease.
Time from entry to exit either by progression or death from prostate cancer stage m0CRPC | 11 years
  M0CRPC as defined by date for clinical assessment of CRPC (Castration Resistant Prostate Cancer) or PSA (Prostate-Specific Antigen) progression ((while on GnRH (Gonadotropin-Releasing Hormone) analogues)) and no date for metastases.
Time from entry to exit either by progression or death from prostate cancer stage m1CRPC | 11 years
  m1CRPC as defined by date for clinical assessment of CRPC or PSA progression (while on GnRH analogues) and confirmed by date for radiographic progression or initiation of treatment for mCRPC (metastatic castration-resistant prostate cancer).
9785-MA-3631: Time from entry to exit either by progression or death from prostate cancer stage m1HSPC | 3.5 years
  M1HSPC as defined by date for start of ADT (bicalutamide or hormone therapy) and date for metastatic disease.
9785-MA-3631: Time from entry to exit either by progression or death from prostate cancer stage m1CRPC | 3.5 years
  M1CRPC as defined by date for clinical assessment of CRPC or PSA progression (while on GnRH analogues) and confirmed by date for radiographic progression or initiation of treatment for mCRPC (metastatic castration-resistant prostate cancer).

SECONDARY OUTCOMES:
Co-morbidities at disease stage m0HSPC | 11 years
  The prevalence of different co-morbidities of interest will be summarized for each disease stage.
Co-morbidities at disease stage m1HSPC | 11 years
  The prevalence of different co-morbidities of interest will be summarized for each disease stage.
Co-morbidities at disease stage m0CRPC | 11 years
  The prevalence of different co-morbidities of interest will be summarized for each disease stage.
Co-morbidities at disease stage m1CRPC | 11 years
  The prevalence of different co-morbidities of interest will be summarized for each disease stage.
Co-medications at disease stage m0HSPC as recorded in the registries | 11 years
  The prevalence of different co-medications of interest will be summarized for each disease stage.
Co-medications at disease stage m1HSPC as recorded in the registries | 11 years
  The prevalence of different co-medications of interest will be summarized for each disease stage.
Co-medications at disease stage m0CRPC as recorded in the registries | 11 years
  The prevalence of different co-medications of interest will be summarized for each disease stage.
Co-medications at disease stage m1CRPC as recorded in the registries | 11 years
  The prevalence of different co-medications of interest will be summarized for each disease stage.
Healthcare resource utilization and related costs in disease stage m0HSPC as measured by number of prostate cancer treatment regimens | 11 years
  Healthcare resource utilization and related costs for each disease stage will be assessed by number of prostate cancer treatment regimens.
Healthcare resource utilization and related costs in disease stage m1HSPC as measured by number of prostate cancer treatment regimens | 11 years
  Healthcare resource utilization and related costs for each disease stage will be assessed by number of prostate cancer treatment regimens.
Healthcare resource utilization and related costs in disease stage m0CRPC as measured by number of prostate cancer treatment regimens | 11 years
  Healthcare resource utilization and related costs for each disease stage will be assessed by number of prostate cancer treatment regimens.
Healthcare resource utilization and related costs in disease stage m1CRPC as measured by number of prostate cancer treatment regimens | 11 years
  Healthcare resource utilization and related costs for each disease stage will be assessed by number of prostate cancer treatment regimens.
Healthcare resource utilization and related costs in disease stage m0HSPC as measured by type of prostate cancer treatment regimens | 11 years
  Healthcare resource utilization and related costs for each disease stage will be assessed by type of prostate cancer treatment regimens.
Healthcare resource utilization and related costs in disease stage m1HSPC as measured by type of prostate cancer treatment regimens | 11 years
  Healthcare resource utilization and related costs for each disease stage will be assessed by type of prostate cancer treatment regimens.
Healthcare resource utilization and related costs in disease stage m0CRPC as measured by type of prostate cancer treatment regimens | 11 years
  Healthcare resource utilization and related costs for each disease stage will be assessed by type of prostate cancer treatment regimens.
Healthcare resource utilization and related costs in disease stage m1CRPC as measured by type of prostate cancer treatment regimens | 11 years
  Healthcare resource utilization and related costs for each disease stage will be assessed by type of prostate cancer treatment regimens.
Healthcare resource utilization and related costs in disease stage m0HSPC as measured by hospitalization in-patient | 11 years
  Healthcare resource utilization and related costs will be assessed by hospitalization in-patient. Disease coding is according to International Classification of Diseases 10th Edition (ICD-10).
Healthcare resource utilization and related costs in disease stage m1HSPC as measured by hospitalization in-patient | 11 years
  Healthcare resource utilization and related costs will be assessed by hospitalization in-patient. Disease coding is according to International Classification of Diseases 10th Edition (ICD-10).
Healthcare resource utilization and related costs in disease stage m0CRPC as measured by hospitalization in-patient | 11 years
  Healthcare resource utilization and related costs will be assessed by hospitalization in-patient. Disease coding is according to International Classification of Diseases 10th Edition (ICD-10).
Healthcare resource utilization and related costs in disease stage m1CRPC as measured by hospitalization in-patient | 11 years
  Healthcare resource utilization and related costs will be assessed by hospitalization in-patient. Disease coding is according to International Classification of Diseases 10th Edition (ICD-10).
Healthcare resource utilization and related costs in disease stage m0HSPC as measured by hospitalization frequency | 11 years
  Healthcare resource utilization and related costs will be assessed by hospitalization frequency. Disease coding is according to International Classification of Diseases 10th Edition (ICD-10).
Healthcare resource utilization and related costs in disease stage m1HSPC as measured by hospitalization frequency | 11 years
  Healthcare resource utilization and related costs will be assessed by hospitalization frequency. Disease coding is according to International Classification of Diseases 10th Edition (ICD-10).
Healthcare resource utilization and related costs in disease stage m0CRPC as measured by hospitalization frequency | 11 years
  Healthcare resource utilization and related costs will be assessed by hospitalization frequency. Disease coding is according to International Classification of Diseases 10th Edition (ICD-10).
Healthcare resource utilization and related costs in disease stage m1CRPC as measured by hospitalization frequency | 11 years
  Healthcare resource utilization and related costs will be assessed by hospitalization frequency. Disease coding is according to International Classification of Diseases 10th Edition (ICD-10).
Healthcare resource utilization and related costs in disease stage m0HSPC as measured by hospitalization duration | 11 years
  Healthcare resource utilization and related costs will be assessed by hospitalization duration. Disease coding is according to International Classification of Diseases 10th Edition (ICD-10).
Healthcare resource utilization and related costs in disease stage m1HSPC as measured by hospitalization duration | 11 years
  Healthcare resource utilization and related costs will be assessed by hospitalization duration. Disease coding is according to International Classification of Diseases 10th Edition (ICD-10).
Healthcare resource utilization and related costs in disease stage m0CRPC as measured by hospitalization duration | 11 years
  Healthcare resource utilization and related costs will be assessed by hospitalization duration. Disease coding is according to International Classification of Diseases 10th Edition (ICD-10).
Healthcare resource utilization and related costs in disease stage m1CRPC as measured by hospitalization duration | 11 years
  Healthcare resource utilization and related costs will be assessed by hospitalization duration. Disease coding is according to International Classification of Diseases 10th Edition (ICD-10).
Healthcare resource utilization and related costs in disease stage m0HSPC as measured by type of hospital visits | 11 years
  Healthcare resource utilization and related costs will be assessed by type of hospital visits.
Healthcare resource utilization and related costs in disease stage m1HSPC as measured by type of hospital visits | 11 years
  Healthcare resource utilization and related costs will be assessed by type of hospital visits.
Healthcare resource utilization and related costs in disease stage m0CRPC as measured by type of hospital visits | 11 years
  Healthcare resource utilization and related costs will be assessed by type of hospital visits.
Healthcare resource utilization and related costs in disease stage m1CRPC as measured by type of hospital visits | 11 years
  Healthcare resource utilization and related costs will be assessed by type of hospital visits.
Healthcare resource utilization and related costs in disease stage m0HSPC as measured by frequency of hospital visits | 11 years
  Healthcare resource utilization and related costs will be assessed by frequency of hospital visits.
Healthcare resource utilization and related costs in disease stage m1HSPC as measured by frequency of hospital visits | 11 years
  Healthcare resource utilization and related costs will be assessed by frequency of hospital visits.
Healthcare resource utilization and related costs in disease stage m0CRPC as measured by frequency of hospital visits | 11 years
  Healthcare resource utilization and related costs will be assessed by frequency of hospital visits.
Healthcare resource utilization and related costs in disease stage m1CRPC as measured by frequency of hospital visits | 11 years
  Healthcare resource utilization and related costs will be assessed by frequency of hospital visits.
Healthcare resource utilization and related costs in disease stage m0HSPC as measured by type of imaging examinations | 11 years
  Healthcare resource utilization and related costs will be assessed by type of imaging examinations.
Healthcare resource utilization and related costs in disease stage m1HSPC as measured by type of imaging examinations | 11 years
  Healthcare resource utilization and related costs will be assessed by type of imaging examinations.
Healthcare resource utilization and related costs in disease stage m0CRPC as measured by type of imaging examinations | 11 years
  Healthcare resource utilization and related costs will be assessed by type of imaging examinations.
Healthcare resource utilization and related costs in disease stage m1CRPC as measured by type of imaging examinations | 11 years
  Healthcare resource utilization and related costs will be assessed by type of imaging examinations.
Healthcare resource utilization and related costs in disease stage m0HSPC as measured by frequency of imaging examinations | 11 years
  Healthcare resource utilization and related costs will be assessed by frequency of imaging examinations.
Healthcare resource utilization and related costs in disease stage m1HSPC as measured by frequency of imaging examinations | 11 years
  Healthcare resource utilization and related costs will be assessed by frequency of imaging examinations.
Healthcare resource utilization and related costs in disease stage m0CRPC as measured by frequency of imaging examinations | 11 years
  Healthcare resource utilization and related costs will be assessed by frequency of imaging examinations.
Healthcare resource utilization and related costs in disease stage m1CRPC as measured by frequency of imaging examinations | 11 years
  Healthcare resource utilization and related costs will be assessed by frequency of imaging examinations.
Healthcare resource utilization and related costs in disease stage m0HSPC as measured by type of laboratory tests | 11 years
  Healthcare resource utilization and related costs will be assessed by type of laboratory tests.
Healthcare resource utilization and related costs in disease stage m1HSPC as measured by type of laboratory tests | 11 years
  Healthcare resource utilization and related costs will be assessed by type of laboratory tests.
Healthcare resource utilization and related costs in disease stage m0CRPC as measured by type of laboratory tests | 11 years
  Healthcare resource utilization and related costs will be assessed by type of laboratory tests.
Healthcare resource utilization and related costs in disease stage m1CRPC as measured by type of laboratory tests | 11 years
  Healthcare resource utilization and related costs will be assessed by type of laboratory tests.
Healthcare resource utilization and related costs in disease stage m0HSPC as measured by frequency of laboratory tests | 11 years
  Healthcare resource utilization and related costs will be assessed by frequency of laboratory tests
Healthcare resource utilization and related costs in disease stage m1HSPC as measured by frequency of laboratory tests | 11 years
  Healthcare resource utilization and related costs will be assessed by frequency of laboratory tests.
Healthcare resource utilization and related costs in disease stage m0CRPC as measured by frequency of laboratory tests | 11 years
  Healthcare resource utilization and related costs will be assessed by frequency of laboratory tests.
Healthcare resource utilization and related costs in disease stage m1CRPC as measured by frequency of laboratory tests | 11 years
  Healthcare resource utilization and related costs will be assessed by frequency of laboratory tests.
9785-MA-3631: Co-morbidities at disease stage m0HSPC | 3.5 years
  The prevalence of different co-morbidities of interest will be summarized for each disease stage.
9785-MA-3631: Co-morbidities at disease stage m1HSPC | 3.5 years
  The prevalence of different co-morbidities of interest will be summarized for each disease stage.
9785-MA-3631: Co-morbidities at disease stage m0CRPC | 3.5 years
  The prevalence of different co-morbidities of interest will be summarized for each disease stage.
9785-MA-3631: Co-morbidities at disease stage m1CRPC | 3.5 years
  The prevalence of different co-morbidities of interest will be summarized for each disease stage.
9785-MA-3631: Co-medications at disease stage m0HSPC as recorded in the registries | 3.5 years
  The prevalence of different co-medications of interest will be summarized for each disease stage.
9785-MA-3631: Co-medications at disease stage m1HSPC as recorded in the registries | 3.5 years
  The prevalence of different co-medications of interest will be summarized for each disease stage.
9785-MA-3631: Co-medications at disease stage m0CRPC as recorded in the registries | 3.5 years
  The prevalence of different co-medications of interest will be summarized for each disease stage.
9785-MA-3631: Co-medications at disease stage m1CRPC as recorded in the registries | 3.5 years
  The prevalence of different co-medications of interest will be summarized for each disease stage.
9785-MA-3631: Prostate Cancer (PCa) treatments for the m1HSPC disease state | 3.5 years
  PCa treatments collected (using real world data) in the m1HSPC population.

CONTACTS AND LOCATIONS:
Overall Officials: Astellas Pharma Europe Ltd., Study Director — Astellas Pharma Europe Ltd.
Locations (1):
- Site SE46001, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=347